CLINICAL TRIAL: NCT04734717
Title: Coordination and Locomotor Problems in Patients With Covid-19 Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Dr. József Tollár, Head of Neurorehabilitation ,7400 Kaposvár, Tallián Gy. u 20-32, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB2021/02
Record Dates: First submitted 2021-02-01; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Motility Disorder; Balance
Keywords: 6MWT; Berg balance; Beam Walking
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID19 (Experimental)
  Interventions: Diagnostic Test: Neurology test
- Controll (Experimental)
  Interventions: Diagnostic Test: Neurology test

INTERVENTIONS:
Diagnostic Test: Neurology test — movement examination of patients with covid19 disease

SUMMARY:
Coordination and Locomotor Problems in Patients With Covid-19 Virus

ELIGIBILITY:
Inclusion Criteria:

* COVID 19 diagnosis

Exclusion Criteria:

* Severe heart problems
* severe demeanor
* alcoholism
* drug problems

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-04-12 (Estimated); Study Completion 2021-04-12 (Estimated)

PRIMARY OUTCOMES:
EQ5D-5L | 5 weeks-long
  Questionnaire
Berg test | 5 weeks-long
  Fatigue questionnaire
SPPB test (gait, balance, leg stregth) | 5 weeks-long
  Walking and balance testing
6MWT | 5 weeks-long
  Walking test

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. József Tollár, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/?term=covid+19+cordination